CLINICAL TRIAL: NCT04499924
Title: A Randomized, Double-blind, Placebo-controlled, Active Comparator Phase 2/3 Study of Tucatinib in Combination With Trastuzumab, Ramucirumab, and Paclitaxel in Subjects With Previously Treated, Locally-advanced Unresectable or Metastatic HER2+ Gastric or Gastroesophageal Junction Adenocarcinoma (GEC)
Brief Title: Tucatinib, Trastuzumab, Ramucirumab, and Paclitaxel Versus Paclitaxel and Ramucirumab in Previously Treated HER2+ Gastroesophageal Cancer
Acronym: MOUNTAINEER-02
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGNTUC-022; C4251004 (Other: Pfizer)
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Results first posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2024-12

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma; Esophageal Adenocarcinoma
Keywords: HER2+; HER2-positive; GEA; GEC; GEJ; Seattle Genetics
MeSH Terms: conditions — Adenocarcinoma Of Esophagus | interventions — tucatinib; Trastuzumab; Ramucirumab; Paclitaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2 Arm (Experimental): Tucatinib + trastuzumab + ramucirumab + paclitaxel
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: ramucirumab; Drug: paclitaxel
- Arm 3A (Experimental): Tucatinib + trastuzumab + ramucirumab + paclitaxel
  Interventions: Drug: tucatinib; Drug: trastuzumab; Drug: ramucirumab; Drug: paclitaxel
- Arm 3B (Active Comparator): Ramucirumab + paclitaxel + tucatinib placebo + trastuzumab placebo
  Interventions: Drug: ramucirumab; Drug: paclitaxel; Other: tucatinib placebo; Other: trastuzumab placebo
- Arm 3C (Experimental): Tucatinib + ramucirumab + paclitaxel + trastuzumab placebo
  Interventions: Drug: tucatinib; Drug: ramucirumab; Drug: paclitaxel; Other: trastuzumab placebo

INTERVENTIONS:
Drug: tucatinib — 300 mg given twice daily orally
  Other Names: TUKYSA, ONT-380, ARRY-380
  Arms: Arm 3A; Arm 3C; Phase 2 Arm
Drug: trastuzumab — 6 mg/kg loading dose will be administered intravenously (IV; into the vein) on Cycle 1 Day 1, followed by 4 mg/kg IV on Cycle 1 Day 15 and then Days 1 and 15 of each cycle thereafter
  Arms: Arm 3A; Phase 2 Arm
Drug: ramucirumab — 8 mg/kg will be administered IV on Days 1 and 15 of each cycle
  Other Names: CYRAMZA
Drug: paclitaxel — 60 or 80 mg/m^2 IV on Days 1, 8, and 15 of each cycle
Other: tucatinib placebo — Given twice daily orally
  Arms: Arm 3B
Other: trastuzumab placebo — IV on Days 1 and 15 of each cycle
  Arms: Arm 3B; Arm 3C

SUMMARY:
This study is being done to see if tucatinib with trastuzumab, ramucirumab and paclitaxel works better than ramucirumab and paclitaxel to treat HER2-positive (HER2+) cancer of the gut (stomach or gastroesophageal cancer). This study will also look at what side effects happen when participants take this combination of drugs. A side effect is anything the drug does other than treating cancer.

Study treatment will be given in 28-day cycles.

In the Phase 2 part of the trial, participants and their doctors will know what drugs are being given (open-label). In the Phase 3 part, the study is "blinded." This means that participants, their doctor, and the study sponsor will not know which drugs are being given.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of locally-advanced unresectable or metastatic HER2+ gastric or gastroesophageal junction adenocarcinoma (GEC)
* HER2+ disease documented since progression of the most recent line of systemic therapy, as follows:

  * Phase 2 paclitaxel dose optimization stage:

    * HER2 amplification in a blood-based NGS assay performed at a central laboratory, or
    * HER2 overexpression/amplification immunohistochemistry (IHC) and in situ hybridization (ISH) (IHC3+ or IHC2+/ISH+) assay of a tumor tissue sample
  * Phase 2 dose expansion stage:

    * Cohort 2A: HER2 amplification in a blood-based NGS assay performed at a central laboratory
    * Cohort 2B: No HER2 amplification by blood-based NGS assay, but HER2 overexpression/amplification by IHC and ISH (IHC3+ or IHC2+/ISH+) assay of a tumor tissue sample
  * Phase 3: HER2 amplification in a blood-based NGS assay performed at a central laboratory
* History of prior treatment with a HER2-directed antibody
* Progressive disease during or after first-line therapy for locally-advanced unresectable or metastatic GEC
* Phase 2: Measurable disease according to RECIST version 1.1
* Phase 3: Measurable or non-measurable disease according to RECIST version 1.1
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Life expectancy of at least 3 months, in the opinion of the investigator

Exclusion Criteria:

* Subjects with squamous cell or undifferentiated GEC
* Having received more than 1 line of prior systemic therapy for locally-advanced unresectable or metastatic disease
* Having received taxanes ≤12 months prior to enrollment, prior treatment with ramucirumab, or prior treatment with tucatinib, lapatinib, neratinib, afatinib, or any other investigational anti-HER2 and/or anti-EGFR tyrosine kinase inhibitor, or with T-DM1, T-Dxd, or any other HER2-directed antibody-drug conjugate
* Phase 2 paclitaxel dose optimization stage only: history of prior partial or total gastrectomy
* Unable to swallow pills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-03-22 (Actual); Primary Completion 2024-04-17 (Actual); Study Completion 2024-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: JoAl Mayor, PharmD, BCOP, Study Director — Seagen Inc.; Michelle Ubowski, PharmD, Study Director — Seagen Inc.
Locations (48):
- United States (30):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Mayo Clinic Arizona, Phoenix, Arizona
  - Arizona Cancer Center / University of Arizona, Tucson, Arizona
  - City of Hope National Medical Center, Duarte, California
  - UCLA Medical Center / David Geffen School of Medicine, Santa Monica, California
  - Rocky Mountain Cancer Centers - Aurora, Aurora, Colorado
  - Cancer Centers of Colorado - Denver, Denver, Colorado
  - SCL Health - St. Mary's Hospital & Medical Center, Grand Junction, Colorado
  - SCL Health Good Samaritan Medical Center Cancer Centers of Colorado, Lafayette, Colorado
  - Lutheran Medical Center - Cancer Centers of Colorado, Wheat Ridge, Colorado
  - Lombardi Cancer Center / Georgetown University Medical Center, Washington D.C., District of Columbia
  - University of Chicago Medical Center, Chicago, Illinois
  - Holden Comprehensive Cancer Center / University of Iowa, Iowa City, Iowa
  - Norton Cancer Institute, Louisville, Kentucky
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Minnesota Oncology Hematology P.A., Saint Paul, Minnesota
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - Roswell Park Cancer Institute, Buffalo, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic - Taussig Cancer Institute, Cleveland, Ohio
  - Oncology Associates of Oregon, Eugene, Oregon
  - University of Pennsylvania / Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Tennessee, Knoxville, Tennessee
  - Tennessee Oncology-Nashville/Sarah Cannon Research Institute, Nashville, Tennessee
  - Texas Oncology - Baylor Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - San Antonio Medical Center, San Antonio, Texas
  - Texas Oncology - Tyler, Tyler, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
- Australia (2):
  - Central Coast Local Health District (Gosford and Wyong Hospitals), Gosford
  - Austin Health, Heidelberg
- Canada (3):
  - London Regional Cancer Program, London Health Sciences Centre, London, Ontario
  - Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - McGill University Department of Oncology / McGill University Health Centre, Montreal, Quebec
- South Korea (8):
  - Dong-A University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center - Oncology, Seoul
  - Samsung Medical Center, Seoul
  - Ajou University Hospital, Suwon
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (2):
  - Sarah Cannon Research Institute UK, London
  - The Christie NHS Foundation Trust, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with locally-advanced unresectable or metastatic human epidermal growth factor receptor 2 positive (HER2+) gastric or gastroesophageal junction adenocarcinoma (GEC) who had received prior treatment with a HER2-directed antibody, and had received 1 prior line of therapy in the advanced disease setting were included in the study. A total of 17 participants were enrolled and treated in the study.
Pre-assignment Details: "Study termination by sponsor" was used as an end of study reason because long-term follow-up was discontinued following the decision to close enrollment. The study status is listed as completed as participants were permitted to receive treatment until they met protocol defined reasons to stop. After treatment discontinuation, participants were followed through the duration of the safety reporting period, and then ended study as no further disease or survival follow-up was required.
Groups:
- Paclitaxel 60 mg/m^2: Participants received paclitaxel 60 milligram per meter square (mg/m^2) intravenously (IV) on Days 1, 8, and 15 of each 28-day cycle, in combination with tucatinib 300 mg orally twice daily (BID), trastuzumab 6 milligram per kilogram (mg/kg) IV loading dose on Cycle 1 Day 1, 4 mg/kg IV dose on Cycle 1 Day 15 and on Days 1 and 15 of each Cycle thereafter, and ramucirumab 8 mg/kg IV on Days 1 and 15. Participants received treatment until unacceptable toxicity, disease progression, withdrawal of consent, or study closure.
- Paclitaxel 80 mg/m^2: Participants received paclitaxel 80 mg/m^2 IV on Days 1, 8, and 15 of each 28-day Cycle, in combination with tucatinib 300 mg orally BID, trastuzumab 6 mg/kg IV loading dose on Cycle 1 Day 1, 4 mg/kg IV dose on Cycle 1 Day 15 and on Days 1 and 15 of each Cycle thereafter, and ramucirumab 8 mg/kg IV on Days 1 and 15. Participants received treatment until unacceptable toxicity, disease progression, withdrawal of consent, or study closure.
Period: Overall Study
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Started | 8 | 9
Completed | 3 | 0
Not Completed | 5 | 9
Not completed — Study termination by sponsor | 4 | 6
Not completed — Withdrawal by Subject | 1 | 3

BASELINE CHARACTERISTICS:
Population: The full analysis set included all participants who received any amount of any study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2 | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.6 (9.5) | 57.6 (8.9) | 55.7 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 9 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 5 | 4 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 5 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicities (DLT) During the First Cycle of Treatment
Description: DLTs were adverse events (AEs), laboratory abnormalities, or treatment modifications that occurred during the first cycle of treatment in the Phase 2 paclitaxel dose optimization stage that were related to paclitaxel, to tucatinib, or to the combination of tucatinib, trastuzumab, ramucirumab and paclitaxel and that met any of the study protocol specified criteria. The relationship of AEs to study drugs was determined by the investigator. AEs that were attributed only to trastuzumab and/or ramucirumab, but not tucatinib or paclitaxel were not considered DLTs.
Time Frame: Cycle 1 (28 days)
Population: The safety analysis set included all participants who received any amount of any study drug. Participants were considered evaluable for DLT if they received at least 75 percent (%) of the planned administrations of each study drug and were followed for at least 1 cycle or if they experienced a DLT during the first cycle.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Participants | 0 | 2

2. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE was any untoward medical occurrence in a participant or clinical investigational participant administered a medicinal product and which did not necessarily have a causal relationship with this treatment. AEs were defined as treatment emergent if they were newly occurring or worsened following study treatment. A TEAE was defined as a newly occurring or worsening AE after the first dose of study treatment (tucatinib, trastuzumab, ramucirumab, or paclitaxel) and up to 30 days after the last dose of study treatment (tucatinib, trastuzumab, ramucirumab, or paclitaxel, whichever was later).
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment (maximum treatment duration= 19.8 months, maximum follow-up duration up to 20.8 months)
Population: The safety analysis set included all participants who received any amount of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Participants | 8 | 9

3. Primary Outcome: Number of Participants With Treatment-emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as abnormalities that are new or worsened on or after receiving the first dose of study treatment up to 30 days after the last dose of study treatment. Laboratory abnormalities included: 1) Blood chemistry: alanine aminotransferase increased, albumin decreased, alkaline phosphatase increased, aspartate aminotransferase increased, calcium corrected for albumin decreased, calcium corrected for albumin increased, creatinine increased, glomerular filtration rate estimated decreased, glucose decreased, lactate dehydrogenase increased, magnesium decreased, magnesium increased, potassium decreased, potassium increased, sodium decreased, sodium increased, and total bilirubin increased; 2) Hematological: hemoglobin decreased, leukocytes decreased, lymphocytes decreased, neutrophils decreased, and platelets decreased.
Time Frame: as for outcome 2
Population: The safety analysis set included all participants who received any amount of any study drug. Here, 'Number Analyzed' signifies participants evaluable for the specified rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Participants
  Hemoglobin decreased | 3 | 7
  Leukocytes decreased | 4 | 9
  Lymphocytes decreased: number analyzed (Participants) | 5 | 8
  Lymphocytes decreased | 2 | 8
  Neutrophils decreased | 5 | 7
  Platelets decreased | 1 | 7
  Alanine aminotransferase increased | 5 | 5
  Albumin decreased | 4 | 4
  Alkaline phosphatase increased | 2 | 0
  Aspartate aminotransferase increased | 6 | 4
  Calcium corrected for albumin decreased | 1 | 5
  Calcium corrected for albumin increased | 0 | 2
  Creatinine increased | 3 | 2
  Glomerular filtration rate, estimated decreased: number analyzed (Participants) | 5 | 7
  Glomerular filtration rate, estimated decreased | 0 | 1
  Glucose decreased | 1 | 2
  Lactate dehydrogenase increased | 1 | 5
  Magnesium decreased | 0 | 7
  Magnesium increased | 0 | 1
  Potassium decreased | 1 | 6
  Potassium increased | 1 | 0
  Sodium decreased | 2 | 4
  Sodium increased | 1 | 1
  Total bilirubin increased | 3 | 2

4. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Values
Description: Vital sign examinations included systolic blood pressure (SBP), diastolic blood pressure (DBP), heart rate. Criteria: SBP greater than or equal to (>=) 120 millimeters of mercury (mm Hg) or DBP >= 80 mm Hg; SBP >= 140 mm Hg or DBP >= 90 mm Hg; SBP >= 160 mm Hg or DBP >= 100 mm Hg), heart rate greater than (>) 100 beats per minute (min). Clinical significance in vital signs abnormalities was judged by investigator. In this outcome measure number of participants with at least 1 clinically significant abnormality in any vital sign are reported.
Time Frame: as for outcome 2
Population: The safety analysis set included all participants who received any amount of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Participants
  SBP >= 120 mm Hg or DBP >= 80 mm Hg | 8 | 9
  SBP >= 140 mm Hg or DBP >= 90 mm Hg | 7 | 9
  SBP >= 160 mm Hg or DBP >= 100 mm Hg | 2 | 3
  Heart rate > 100 beats per min | 1 | 4

5. Primary Outcome: Maximum Percentage Change From Baseline in Weight
Description: Maximum percentage decrease from baseline in weight is reported in this outcome measure.
Time Frame: From Baseline (Day 1) up to 30 days after the last dose of study treatment (maximum treatment duration= 19.8 months, maximum follow-up duration up to 20.8 months)
Population: The safety analysis set included all participants who received any amount of any study drug.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Percent Change | 0.34 [-4.3 to 9.9] | 6.21 [-4.8 to 21.0]

6. Primary Outcome: Number of Participants With Any Dose Modifications
Description: Dose modification included dose hold, dose reduction, dose error and unplanned dose adjustments. Number of participants with any dose treatment modifications for paclitaxel, ramucirumab, trastuzumab, and tucatinib are reported in this outcome measure.
Time Frame: From first dose of the study treatment (Day 1) up to the last dose of study treatment (maximum treatment duration up to 19.8 months)
Population: The full analysis set included all participants who received any amount of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Participants
  Paclitaxel | 7 | 9
  Ramucirumab | 7 | 8
  Trastuzumab | 7 | 8
  Tucatinib | 6 | 8

7. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors (RECIST) Version (v) 1.1 By Investigator Assessment
Description: ORR was defined as the percentage of participants with best overall response of complete response (CR) or partial response (PR) according to RECIST v 1.1 by investigator assessment. As per RECIST v1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to less than (<) 10 millimeter (mm). PR was defined as at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. As per RECIST v1.1, disease progression (PD) was defined as one of the following: at least a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) with an absolute increase of at least 5mm, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: From the first dose of study treatment until the first documented CR or PR on or before the first documented PD or new anti-cancer therapies or death, whichever occurred first (up to 19.8 months)
Population: The response evaluable analysis set included all participants who had baseline disease assessment, received study treatment, had post baseline disease assessment or discontinued treatment due to documented disease progression, clinical progression, AEs, or death.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Percentage of participants | 50.0 [15.7 to 84.3] | 100.0 [66.4 to 100.0]

8. Secondary Outcome: Confirmed ORR Per RECIST v1.1 By Investigator Assessment
Description: Confirmed ORR was defined as the percentage of participants with best overall response of confirmed CR or PR according to RECIST v1.1 by investigator assessment. For a response to be confirmed, the subsequent response needs to be at least 4 weeks after the initial response. As per RECIST v1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30 % decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. As per RECIST v1.1, disease progression (PD) was defined as one of the following: at least a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) with an absolute increase of at least 5mm, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions.
Time Frame: From the first dose of study treatment until the first documented confirmed CR or PR or before the first documented PD or new anti-cancer therapies or death, whichever occurred first (up to 19.8 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Percentage of participants | 37.5 [8.5 to 75.5] | 100.0 [66.4 to 100.0]

9. Secondary Outcome: Progression-Free Survival (PFS) Per RECIST v1.1 By Investigator Assessment
Description: PFS was defined as the time from the date of treatment initiation to the date of documented PD or death from any cause, whichever occurred first per RECIST version 1.1 by investigator assessment. As per RECIST v1.1, disease progression (PD) was defined as one of the following: at least a 20% increase in the sum of diameters (SOD) of target lesions (taking as reference the smallest sum on study) with an absolute increase of at least 5mm, unequivocal progression of existing non-target lesions, or the appearance of one or more new lesions. Participants without documentation of PD or death at the time of analysis were censored at the date of the last tumor assessment. Kaplan-Meier method was used for evaluation.
Time Frame: From the date of first dose until the first documentation of PD or death or censoring date, whichever occurred first (up to 19.8 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Months | 4.1 [1.5 to 12.5] | 12.2 [7.0 to 14.4]

10. Secondary Outcome: Duration of Response (DOR) Per RECIST v1.1 By Investigator Assessment
Description: DOR: time from first documentation of objective response of CR or PR to first documentation of PD or death from any cause, whichever occurred first according to RECIST v1.1 by investigator assessment. As per RECIST v1.1, CR: disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10mm. PR: at least a 30% decrease in sum of diameters of target lesions, taking as reference baseline sum diameters. PD was defined as one of the following: at least a 20% increase in sum of diameters of target lesions (taking as reference the smallest sum on study) with an absolute increase of at least 5mm, unequivocal progression of existing non-target lesions, or appearance of one or more new lesions. Participants without documentation of PD or death at time of analysis were censored at the date of last tumor assessment. Kaplan-Meier method was used for evaluation.
Time Frame: From the first documented CR or PR until the first documentation of PD or death or censoring date, whichever occurred first (up to 19.8 months)
Population: The response evaluable analysis set included all participants who had baseline disease assessment, received study treatment, had post baseline disease assessment or discontinued treatment due to documented disease progression, clinical progression, AEs, or death. Here, "Number of Participants Analyzed" signifies participants who had CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 9
Months | 10.6 [2.8 to NA] — Upper limit of 95% CI could not be estimated due to insufficient number of participants with event. | 11.0 [2.9 to 12.9]

11. Secondary Outcome: Disease Control Rate (DCR) Per RECIST v1.1 By Investigator Assessment
Description: DCR was defined as percentage of participants with CR, PR, or stable disease (SD or non-CR/non-progressive disease) according to RECIST v1.1 by investigator assessment. As per RECIST v1.1, CR was defined as disappearance of all target and non-target lesions and normalization of tumor markers. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. PR was defined as at least a 30 % decrease in sum of diameters of target lesions, taking as reference the baseline sum diameters. PD was defined as one of following: at least a 20% increase in the sum of diameters of target lesions (taking as reference the smallest sum on study) with an absolute increase of at least 5mm, unequivocal progression of existing non-target lesions, or appearance of one or more new lesions. SD was defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference smallest sum of diameters.
Time Frame: From the first dose study treatment until PD or death, whichever occurred first (up to 19.8 months)
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Percentage of participants | 87.5 [47.3 to 99.7] | 100.0 [66.4 to 100.0]

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve to the Time of the Last Quantifiable Concentration (AUClast) of Paclitaxel, Tucatinib and Their Metabolites
Description: AUClast was reported for tucatinib, tucatinib metabolite (ONT-993), paclitaxel and paclitaxel metabolites (6 alpha-hydroxy-paclitaxel, 3'-p-hydroxy-paclitaxel and 6 alpha-3'-p-Dihydroxy-paclitaxel).
Time Frame: Tucatinib and ONT-993- Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 2, 4, 6, 8 hours post-dose; Paclitaxel and its metabolites- Cycle 1 Days 1 and 8, Cycle 2 Day 1: Pre-dose, 2, 4, 6, 8 hours post-dose (each cycle length=28 days)
Population: The pharmacokinetics (PK) analysis set included participants in the full analysis set who received at least one dose of tucatinib or paclitaxel and have at least one evaluable PK assessment. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Hour*nanograms per milliliter
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Hour*nanograms per milliliter
  Cycle 1 Day 8: Tucatinib: number analyzed (Participants) | 5 | 7
  Cycle 1 Day 8: Tucatinib | 4210 (37.7) | 3210 (60.0)
  Cycle 1 Day 8: ONT-993: number analyzed (Participants) | 5 | 7
  Cycle 1 Day 8: ONT-993 | 550 (65.3) | 521 (92.1)
  Cycle 2 Day 1: Tucatinib: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: Tucatinib | 2810 (34.7) | 3130 (35.8)
  Cycle 2 Day 1: ONT-993: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: ONT-993 | 348 (10.1) | 423 (50.4)
  Cycle 1 Day 1: Paclitaxel: number analyzed (Participants) | 7 | 6
  Cycle 1 Day 1: Paclitaxel | 2180 (45.5) | 3500 (10.1)
  Cycle 1 Day 1: 6 alpha-hydroxy-paclitaxel: number analyzed (Participants) | 7 | 6
  Cycle 1 Day 1: 6 alpha-hydroxy-paclitaxel | 118 (117) | 133 (100)
  Cycle 1 Day 1: 3'-p-hydroxy-paclitaxel: number analyzed (Participants) | 7 | 6
  Cycle 1 Day 1: 3'-p-hydroxy-paclitaxel | 49.7 (123) | 77.8 (40.8)
  Cycle 1 Day 1: 6 alpha-3'-p-dihydroxy-paclitaxel: number analyzed (Participants) | 7 | 4
  Cycle 1 Day 1: 6 alpha-3'-p-dihydroxy-paclitaxel | 38.9 (194) | 42.0 (242)
  Cycle 1 Day 8: Paclitaxel: number analyzed (Participants) | 6 | 7
  Cycle 1 Day 8: Paclitaxel | 2210 (54.6) | 3220 (41.5)
  Cycle 1 Day 8: 6 alpha-hydroxy-paclitaxel: number analyzed (Participants) | 6 | 7
  Cycle 1 Day 8: 6 alpha-hydroxy-paclitaxel | 92.7 (109) | 155 (88.3)
  Cycle 1 Day 8: 3'-p-hydroxy-paclitaxel: number analyzed (Participants) | 6 | 7
  Cycle 1 Day 8: 3'-p-hydroxy-paclitaxel | 11.7 (106) | 24.3 (89.6)
  Cycle 1 Day 8: 6 alpha-3'-p-dihydroxy-paclitaxel: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 8: 6 alpha-3'-p-dihydroxy-paclitaxel | 7.56 (175) | 14.1 (128)
  Cycle 2 Day 1: Paclitaxel: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: Paclitaxel | 2380 (45.9) | 3120 (31.4)
  Cycle 2 Day 1: 6 alpha-hydroxy-paclitaxel: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: 6 alpha-hydroxy-paclitaxel | 51.2 (56.9) | 136 (116)
  Cycle 2 Day 1: 3'-p-hydroxy-paclitaxel: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: 3'-p-hydroxy-paclitaxel | 11.3 (77.0) | 24.5 (97.5)
  Cycle 2 Day 1: 6 alpha-3'-p-dihydroxy-paclitaxel: number analyzed (Participants) | 3 | 5
  Cycle 2 Day 1: 6 alpha-3'-p-dihydroxy-paclitaxel | 5.48 (251) | 12.6 (250)

13. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax)
Description: Cmax was reported for tucatinib and tucatinib metabolite ONT-993.
Time Frame: Tucatinib and ONT-993- Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 2, 4, 6, 8 hours post-dose (each cycle length=28 days)
Population: The PK analysis set included participants in the full analysis set who received at least one dose of tucatinib or paclitaxel and have at least one evaluable PK assessment. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed" signifies participants evaluable for the specified rows.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Nanograms per milliliter (ng/mL)
  Cycle 1 Day 8: Tucatinib: number analyzed (Participants) | 6 | 9
  Cycle 1 Day 8: Tucatinib | 769 (30.9) | 615 (56.1)
  Cycle 2 Day 1: Tucatinib: number analyzed (Participants) | 4 | 8
  Cycle 2 Day 1: Tucatinib | 482 (21.4) | 553 (52.3)
  Cycle 1 Day 8: ONT-993: number analyzed (Participants) | 6 | 9
  Cycle 1 Day 8: ONT-993 | 112 (65.2) | 130 (99.9)
  Cycle 2 Day 1: ONT-993: number analyzed (Participants) | 4 | 8
  Cycle 2 Day 1: ONT-993 | 79.0 (35.7) | 84.2 (80.3)

14. Secondary Outcome: Time to Maximum Observed Plasma Concentration (Tmax)
Description: Tmax was reported for tucatinib and tucatinib metabolite ONT-993.
Time Frame: Tucatinib and ONT-993- Cycle 1 Day 8, Cycle 2 Day 1: Pre-dose, 2, 4, 6, 8 hours post-dose (each cycle length=28 days)
Population: as for outcome 13
Measure: Median (Full Range); unit: Hours
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Hours
  Cycle 1 Day 8: Tucatinib: number analyzed (Participants) | 6 | 9
  Cycle 1 Day 8: Tucatinib | 3.5 [2.0 to 6.6] | 3.9 [1.7 to 7.5]
  Cycle 2 Day 1: Tucatinib: number analyzed (Participants) | 4 | 8
  Cycle 2 Day 1: Tucatinib | 3.0 [1.4 to 4.9] | 3.9 [1.5 to 5.9]
  Cycle 1 Day 8: ONT-993: number analyzed (Participants) | 6 | 9
  Cycle 1 Day 8: ONT-993 | 1.2 [1.0 to 2.2] | 1.9 [1.0 to 3.9]
  Cycle 2 Day 1: ONT-993: number analyzed (Participants) | 4 | 8
  Cycle 2 Day 1: ONT-993 | 1.3 [1.1 to 2.0] | 2.8 [1.1 to 4.0]

15. Secondary Outcome: Trough Concentration (Ctrough)
Description: Ctrough was calculated for tucatinib and tucatinib metabolite ONT-993.
Time Frame: Tucatinib and ONT-993- Cycle 1 Day 8, Cycle 2 Day 1: Predose (each cycle length=28 days)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Nanograms per milliliter (ng/mL)
  Cycle 1 Day 8: Tucatinib: number analyzed (Participants) | 5 | 9
  Cycle 1 Day 8: Tucatinib | 71.0 (2010) | 156 (64.3)
  Cycle 2 Day 1: Tucatinib: number analyzed (Participants) | 6 | 7
  Cycle 2 Day 1: Tucatinib | 67.4 (1180) | 62.0 (1320)
  Cycle 1 Day 8: ONT-993: number analyzed (Participants) | 5 | 9
  Cycle 1 Day 8: ONT-993 | 9.64 (289) | 17.4 (75.7)
  Cycle 2 Day 1: ONT-993: number analyzed (Participants) | 6 | 7
  Cycle 2 Day 1: ONT-993 | 8.23 (203) | 8.45 (251)

16. Secondary Outcome: Metabolite Ratio Based on AUClast (MRAUClast)
Description: MRAUClast was defined as metabolic ratio, that is, ratio of the AUClast of a given paclitaxel metabolite over the AUClast of paclitaxel. MRAUClast for 6 alpha-hydroxypaclitaxel, 3-p-hydroxy-paclitaxel and 6 alpha-3-p-dihydroxy-paclitaxel was reported in this outcome measure.
Time Frame: Paclitaxel and its metabolites- Cycle 1 Days 1 and 8, Cycle 2 Day 1: Pre-dose, 2, 4, 6, 8 hours post-dose (each cycle length=28 days)
Population: The PK analysis set included participants in the full analysis set who received at least one dose of tucatinib or paclitaxel and have at least one evaluable PK assessment. All participants reported under "Number of Participants Analyzed" contributed data to the table; however, may not have evaluable data for every row. Here, "Number Analyzed' signifies participants evaluable for the specified rows. Only non-zero values for each time point have been reported in this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Ratio
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 8 | 9
Ratio
  Cycle 1 Day 1: 6 alpha-hydroxypaclitaxel: number analyzed (Participants) | 7 | 6
  Cycle 1 Day 1: 6 alpha-hydroxypaclitaxel | 0.0532 (92.5) | 0.0373 (104)
  Cycle 1 Day 1: 3-p-hydroxypaclitaxel: number analyzed (Participants) | 7 | 6
  Cycle 1 Day 1: 3-p-hydroxypaclitaxel | 0.0224 (99.4) | 0.0218 (43.0)
  Cycle 1 Day 1: 6 alpha-3-p-dihydroxypaclitaxel: number analyzed (Participants) | 7 | 4
  Cycle 1 Day 1: 6 alpha-3-p-dihydroxypaclitaxel | 0.0172 (151) | 0.0115 (269)
  Cycle 1 Day 8: 6 alpha-hydroxypaclitaxel: number analyzed (Participants) | 6 | 7
  Cycle 1 Day 8: 6 alpha-hydroxypaclitaxel | 0.0412 (67.3) | 0.0474 (130)
  Cycle 1 Day 8: 3-p-hydroxypaclitaxel: number analyzed (Participants) | 6 | 7
  Cycle 1 Day 8: 3-p-hydroxypaclitaxel | 0.00519 (78.3) | 0.00741 (101)
  Cycle 1 Day 8: 6 alpha-3-p-dihydroxypaclitaxel: number analyzed (Participants) | 6 | 6
  Cycle 1 Day 8: 6 alpha-3-p-dihydroxypaclitaxel | 0.00330 (130) | 0.00445 (205)
  Cycle 2 Day 1: 6 alpha-hydroxypaclitaxel: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: 6 alpha-hydroxypaclitaxel | 0.0212 (47.9) | 0.0428 (120)
  Cycle 2 Day 1: 3-p-hydroxypaclitaxel: number analyzed (Participants) | 4 | 7
  Cycle 2 Day 1: 3-p-hydroxypaclitaxel | 0.00467 (33.1) | 0.00772 (78.0)
  Cycle 2 Day 1: 6 alpha-3-p-dihydroxypaclitaxel: number analyzed (Participants) | 3 | 5
  Cycle 2 Day 1: 6 alpha-3-p-dihydroxypaclitaxel | 0.00222 (108) | 0.00340 (304)

ADVERSE EVENTS:
Time Frame: From first dose of the study treatment (Day 1) up to 30 days after the last dose of study treatment (maximum treatment duration= 19.8 months, maximum follow-up duration up to 20.8 months)
Description: Same event may appear as both non-serious adverse event (SAE) and SAE; however, what is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in another participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set was evaluated. All-cause mortality: number of deaths are reported from Day 1 of study up to 30 days post last dose and deaths which occurred after 30 days post last dose of study drug are also included.
Arm/Group | Paclitaxel 60 mg/m^2 | Paclitaxel 80 mg/m^2
All-Cause Mortality (participants affected / at risk) | 3/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 4/8 | 5/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel 60 mg/m^2 (N=8) | Paclitaxel 80 mg/m^2 (N=9)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Intestinal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Paclitaxel 60 mg/m^2 (N=8) | Paclitaxel 80 mg/m^2 (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 (3) | 2 (6)
Neutropenia (Blood and lymphatic system disorders) | 1 (8) | 5 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Tympanic membrane perforation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1)
Ocular hyperaemia (Eye disorders) | 0 (0) | 1 (1)
Photophobia (Eye disorders) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 1 (3)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 2 (5)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 3 (4)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 4 (7)
Diarrhoea (Gastrointestinal disorders) | 4 (8) | 8 (59)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1)
Eructation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gingival oedema (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (3) | 7 (17)
Odynophagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 2 (2) | 5 (5)
Swollen tongue (Gastrointestinal disorders) | 0 (0) | 1 (1)
Tongue haematoma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (8)
Chills (General disorders) | 1 (1) | 1 (2)
Discomfort (General disorders) | 0 (0) | 1 (1)
Face oedema (General disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 2 (2) | 7 (11)
Localised oedema (General disorders) | 1 (1) | 1 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 2 (2)
Pain (General disorders) | 0 (0) | 1 (1)
Peripheral swelling (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 3 (3)
Temperature intolerance (General disorders) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 1 (4)
Hypersensitivity (Immune system disorders) | 0 (0) | 2 (2)
COVID-19 (Infections and infestations) | 1 (1) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (2)
Rectal abscess (Infections and infestations) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 2 (4)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (2)
Hyphaema (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 1 (1) | 2 (5)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Ejection fraction decreased (Investigations) | 2 (3) | 1 (1)
Serum ferritin decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 2 (2) | 4 (4)
Decreased appetite (Metabolism and nutrition disorders) | 1 (2) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 2 (2)
Dysgeusia (Nervous system disorders) | 0 (0) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 3 (7)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 7 (9)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 4 (4)
Hallucination (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 3 (3)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Chromaturia (Renal and urinary disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 6 (8)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Paranasal sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (3)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 (3) | 2 (2)
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychomadesis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (5)
Rash (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (5)
Hypotension (Vascular disorders) | 1 (1) | 2 (3)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1)
Peripheral coldness (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Study had following parts: Phase (P)2 (paclitaxel DO (dose optimization), DE (dose expansion)), and P3. P2 DE, and P3 not initiated (sponsor decision). After DO completed enrollment, long-term follow-up discontinued. Participants received treatment until protocol-defined discontinuation criteria met. After treatment discontinued, participants followed through duration of safety period. So, results in all sections reported only for paclitaxel DO (P2) not for DE (P2), and P3.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-02): https://cdn.clinicaltrials.gov/large-docs/24/NCT04499924/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT04499924/SAP_001.pdf